CLINICAL TRIAL: NCT00547872
Title: Screening Asymptomatic Patients With Diabetes for Unknown Coronary Artery Disease: an Open-label Randomized Study Comparing Exercise Testing Strategy With Management Based on Pharmacological/Behavioral Treatment of Traditional Risk Factors
Brief Title: Exercise Testing to Screen for Unknown Coronary Artery Disease in Diabetic Patients: Does it Contribute to a Risk Reduction in Very High Risk Patients?
Acronym: DADDY-D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TURRINI FABRIZIO (Other)
Responsible Party: Sponsor-Investigator, TURRINI FABRIZIO, Turrini fabrizio MD, Azienda Unita' Sanitaria Locale Di Modena
Organization: Azienda Unita' Sanitaria Locale Di Modena (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCV-MO-07-001
Record Dates: First submitted 2007-10-17; First posted 2007-10-23 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Best medical/behavioral treatment according to guidelines suggestions plus CAD screening by ECG tolerance testing followed by revascularization in case of coronary stenosis.
  Interventions: Procedure: exercise testing - coronary angiography - revascularization
- 2 (No Intervention): Best medical/behavioral treatment according to guidelines suggestions

INTERVENTIONS:
Procedure: exercise testing - coronary angiography - revascularization — Those patients with a positive exercise ECG test will be studied by coronary angiography and treated according to the severity of coronary lesions by percutaneous stenting or surgery
  Other Names: Exercise tolerance testing as screening; Coronary angiography; Revascularization surgical or pecutaneous
  Arms: 1

SUMMARY:
In the present study a cohort of diabetic patients without any symptoms and without known coronary artery disease (CAD) will be screened at the investigators' diabetes outpatients services. Those with intermediate or high risk will be asked to participate and enrolled. They will be seen and followed by the cardiologists in order to provide the best adherence to medical therapy. By mean of a randomization process, a group of patients will undergo an exercise electrocardiography (ECG) testing while the other group will continue to be regularly seen at the investigators' cardiology service. Those patients with a positive exercise ECG test will be study by coronary angiography and treated according to the severity of coronary lesions by percutaneous stenting or surgery. Both groups of patients will be seen every six-eight months for the next three years.

ELIGIBILITY:
Inclusion Criteria:

* Type two Diabetes Mellitus
* Cardiovascular risk equal or higher than 10% according to Italian risk score (www.cuore.iss.it)

Exclusion Criteria:

* Known coronary artery disease
* Symptomatic heart failure
* Objective inability to perform treadmill exercise
* Known or active malignancy, advanced renal failure (clearance < 25 ml/mi/1.73m2), liver cirrhosis (child Pugh III); stroke within the past 30 days
* Presence of left bundle branch block or ST depression at rest greater than 0.9 mm

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2007-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Death and myocardial infarction | three years

SECONDARY OUTCOMES:
Symptomatic heart failure | three years

CONTACTS AND LOCATIONS:
Overall Officials: fabrizio turrini, Principal Investigator — Azienda Unità Sanitaria Locale di Modena
Locations (1):
- Nuovo Ospedale Civile Sant'Agostino Estense, Modena, MO, Italy

REFERENCES:
- [Background] Turrini F, Messora R, Giovanardi P, Tondi S, Magnavacchi P, Cavani R, Tosoni G, Cappelli C, Pellegrini E, Romano S, Baldini A, Zennaro RG, Bondi M. Screening asymptomatic patients with diabetes for unknown coronary artery disease: does it reduce risk? An open-label randomized trial comparing a strategy based on exercise testing aimed at revascularization with management based on pharmacological/behavioural treatment of traditional risk factors. DADDY-D Trial (Does coronary Atherosclerosis Deserve to be Diagnosed and treated early in Diabetics?). Trials. 2009 Dec 23;10:119. doi: 10.1186/1745-6215-10-119. PMID 20030830
- [Derived] Turrini F, Scarlini S, Mannucci C, Messora R, Giovanardi P, Magnavacchi P, Cappelli C, Evandri V, Zanasi A, Romano S, Cavani R, Ghidoni I, Tondi S, Bondi M. Does coronary Atherosclerosis Deserve to be Diagnosed earlY in Diabetic patients? The DADDY-D trial. Screening diabetic patients for unknown coronary disease. Eur J Intern Med. 2015 Jul;26(6):407-13. doi: 10.1016/j.ejim.2015.05.006. Epub 2015 Jun 6. PMID 26058988